CLINICAL TRIAL: NCT00841282
Title: Comparison of Study Versus Conventional Method for Performing Colonoscopy by Supervised Trainees for Colorectal Cancer Screening and Surveillance
Brief Title: RCT of Air Insufflation Versus Water Infusion Colonoscopy by Supervised Trainees
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: East Bay Institute for Research and Education (Other)
Responsible Party: Joseph Leung, MD, Section of Gastroenterology, Sacramento VA Medical Center
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: EBIRE-GI-002
Record Dates: First submitted 2009-02-09; First posted 2009-02-11 (Estimated); Last update posted 2009-02-11 (Estimated); Status verified 2009-02

CONDITIONS: Colorectal Cancer
Keywords: Colorectal cancer screening; Optical colonoscopy; Water method; Sedation
MeSH Terms: conditions — Colorectal Neoplasms | interventions — Colonoscopy

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Active Comparator): Water Infusion in lieu of Air Insufflation Colonoscopy
  Interventions: Procedure: Colonoscopy for colorectal cancer screening; Procedure: Water Infusion Colonoscopy
- 2 (Placebo Comparator): Air Insufflation Colonoscopy
  Interventions: Procedure: Colonoscopy for colorectal cancer screening; Procedure: Air insufflation colonoscopy

INTERVENTIONS:
Procedure: Colonoscopy for colorectal cancer screening
Procedure: Water Infusion Colonoscopy — water infusion in lieu of air insufflation for screening colonoscopy
  Arms: 1
Procedure: Air insufflation colonoscopy — Conventional colonoscopy with air insufflation
  Arms: 2

SUMMARY:
Our aim is to perform a randomized-controlled trial comparing air insufflation sedated colonoscopy (conventional method) vs. water infusion sedated colonoscopy (study method) by supervised trainees. Randomized trials demonstrating reduced need for sedation medications without compromising patients' comfort, cecal intubation rates or polyps detection may cause a paradigm shift and positively alter the way traditional colonoscopy is performed and future endoscopists are trained.

DETAILED DESCRIPTION:
Background: A novel water method permitted 52% of patients accepting on-demand sedation to complete colonoscopy without medications and significantly increased successful cecal intubation from 76% to 97% in patients accepting scheduled unsedated colonoscopy.

Aim: To perform a randomized controlled trial comparing air insufflation (conventional method) vs. water infusion in lieu of air (study method) colonoscopy in minimally sedated patients by supervised trainees.

Hypothesis: Compared with the conventional method, patients examined by the study method have lower pain scores and require less medication but have similar cecal intubation rate and willingness to repeat future colonoscopy.

Setting: Outpatient colonoscopy in a single VA hospital Methods: After informed consent and standard bowel preparation, patients received pre-medications administered as 0.5 increment of Fentanyl (25 μg) and 0.5 increment of Versed (1 mg) plus 50 mg Diphenhydramine. The conventional and the study method for colonoscopy were implemented as previously described. Additional pain medications were administered at the patients' request.

Outcome measures: Increments of medications, pain scores, cecal intubation and willingness to repeat colonoscopy.

Limitations: Single VA site, older male population

ELIGIBILITY:
Inclusion criteria:

* Adult (> 50 years old) male and female patients who are scheduled and consented for screening or surveillance colonoscopy,
* Accept randomization to the study or the conventional method, and agree to complete study questionnaires
* The adults will be normal healthy patients or patients with mild systemic disease, ASA 1 or ASA 2

Exclusion criteria:

* Patients who have contraindications for sedation, decline to participate, unable to give informed consent or complete the questionnaires due to language or other difficulties will be excluded
* Excluded patients will be managed by usual procedures

Ages: 50 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 62 (Actual)
Dates: Start 2008-10; Primary Completion 2009-02 (Actual); Study Completion 2009-02 (Actual)

PRIMARY OUTCOMES:
Increments of medications used for sedation | duration of procedure

SECONDARY OUTCOMES:
pain score during colonoscopy | duration of procedure
success of cecal intubation | duration of study
willingness to repeat colonoscopy | duration of study

CONTACTS AND LOCATIONS:
Locations (1):
- Sacramento VA Medical Center,, Mather, California, United States